CLINICAL TRIAL: NCT03927352
Title: A Phase 3, Randomized, Double-blind Study Evaluating the Efficacy and Safety of SCT630 Compared With Adalimumab in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: The Purpose of This Research Study is to Compare the Efficacy and Safety of SCT630 and Adalimumab (HUMIRA®) in Adults With Plaque Psoriasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCT630PS03
Record Dates: First submitted 2019-04-22; First posted 2019-04-25 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT630 (Experimental): Participants received 80 mg SCT630 subcutaneously on week 1/day 1 (initial loading dose) and 40 mg at week 2 and every 2 weeks thereafter until week 16.
  Participants with a PASI 50 response at week 16 continued to receive 40 mg SCT630 until week 48.
  Interventions: Biological: SCT630
- adalimumab-EU source (Active Comparator): Participants received 80 mg adalimumab subcutaneously on week 1/day 1 (initial loading dose) and 40 mg at week 2 and every 2 weeks thereafter until week 16.
  At week 16 participants with a PASI 50 response were re-randomized to treatment with adalimumab or were transitioned to SCT630 until week 48
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: SCT630 — Administered by subcutaneous injection
  Arms: SCT630
Biological: Adalimumab — Administered by subcutaneous injection
  Arms: adalimumab-EU source

SUMMARY:
The purpose of this research study is to compare the efficacy and safety of SCT630 and adalimumab (HUMIRA®) in adults with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 and ≤ 70 years of age at time of screening.
2. History of psoriasis for at least 6 months ,and stable moderate to severe plaque psoriasis within 2 months prior to randomized.
3. Moderate to severe psoriasis defined at screening and baseline by：Body surface area (BSA) affected by plaque psoriasis of 10% or greater, and PASI score of 12 or greater, and static physician's global assessment score of 3 or greater.
4. Negative test for Interferon-gamma-release assay an chest X-ray at time of screening.
5. Subject is a candidate for systemic therapy or phototherapy procedures.
6. Female participants must have a negative pregnancy test; are not planning to become pregnant; and must not be lactating.
7. From the screening period to the end (Six months after the last administration),female participants must agree to employ a highly effective contraceptive measure.

Exclusion Criteria:

1. Other forms of psoriasis,skin conditions(eg, eczema) or systemic autoimmune diseases which affected the evaluation of treatment outcomes .
2. Received local anti-psoriasis drugs within 2weeks prior to baseline;
3. Received PUVA ,UVB or non-biologics within 4weeks prior to baseline,including methotrexate,Cyclosporine,tretinoins,traditional Chinese medicine,and so on.
4. Received etanercept or its biosimilars within 4weeks prior to baseline.
5. Received other anti-TNF ,IL-12/23inhibitors or IL-17inhibitors within12months prior to baseline.
6. Be receiving or had received any biologics ≤ five half-lives.
7. Patients who previously used adalimumab or a biosimilar of adalimumab ineffectively or intolerantly.
8. History of tuberculosis, active tuberculosis or latent tuberculosis infection.
9. Suffering from active infection or history of infection :Systemic anti-infective therapy was performed 4 weeks before screening, severe infections with hospitalization or intravenous anti-infective treatment within 8 weeks before screening or recurrent, chronic or other active infections which were assessed by researchers to increase the risk of subjects.
10. Subjects were known to have malignant tumors or a history of malignant tumors (except for skin squamous cell carcinoma in situ, basal cell carcinoma, cervical cancer in situ, or skin squamous cell carcinoma with no evidence of recurrence after thorough treatment, or five years prior to investigational product administration)
11. Moderate to severe congestive heart failure (New York Heart Association Classes III or IV）.
12. Subjects with a significant disease other than psoriasis and/or a significant uncontrolled disease (such as, but not limited to, nervous system, renal, hepatic, endocrine, hematological, autoimmune or gastrointestinal disorders)，and which were assessed by researchers to increase the risk of subjects.
13. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times upper limit of normal (ULN) ,Hemoglobin < 90 g/L ,Leukocyte count < 3.5×109/L,Platelets < 100×109/L ,Serum creatinine > 2.5 times upper limit of normal (ULN) at Screening.
14. Received any live vaccines ≤4 weeks prior to investigational product administration,or patients who are expecting to receive any live vaccines during the trial.
15. Subjects had hypersensitivity to test drugs and their excipients, or drugs with the same pharmacological and biological classification as test drugs, and had a history of allergy to active substances or excipients of adalimumab or SCT630.
16. Positive test for anti-nuclear antibody(ANA) or anti-double-stranded DNA antibody at screening.
17. Subjects were accompanied by active neuropathy, including but not limited to multiple sclerosis, Guillain-Barre syndrome, optic neuritis, transverse myelitis, or neurological symptoms suggesting demyelinating lesions of the central nervous system.
18. Positive test for HIV antibodies, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies ,or Treponema pallidum antibody at screening.
19. The results of five tests for hepatitis B virus infection should be further tested for hepatitis B virus DNA, if it is greater than or equal to the upper limit of the reference value of each hospital.
20. Women who are pregnant or nursing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent Improvement From Baseline in Psoriasis Area and Severity Index (PASI) at Week 16 | Baseline and Week 16
  The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
  Percent improvement from baseline was calculated as (value at baseline - value at post-baseline visit) × 100 / (value at baseline).

SECONDARY OUTCOMES:
Percent Improvement From Baseline in PASI at Week 4、8、12、24、32、48、50 | Baseline and week 4、8、12、24、32、48、50
  The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
  Percent improvement from baseline is calculated as (value at baseline - value at post-baseline visit) × 100 / (value at baseline).
Percentage of Participants With a PASI 75 Response at Week 4、8、12、16、24、32、48、50 | Baseline and Week 4、8、12、16、24、32、48、50
  A PASI 75 response is a 75% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Percentage of Participants With a PASI 50 Response at Week 4、8、12、16、24、32、48、50 | Baseline and Week 4、8、12、16、24、32、48、50
  A PASI 50 response is a 50% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Percentage of Participants With a PASI 90 Response at Week 4、8、12、16、24、32、48、50 | Baseline and Week 4、8、12、16、24、32、48、50
  A PASI 90 response is a 90% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Percentage of Participants With a PASI 100 Response at Week 4、8、12、16、24、32、48、50 | Baseline and Week 4、8、12、16、24、32、48、50
  A PASI 100 response is a 100% or greater improvement (reduction) from baseline in PASI score. The PASI measures the average redness (erythema), thickness (induration), and scaliness (each graded on a 0 to 4 scale) of psoriasis lesions, weighted by the area of involvement in the four main body areas (i.e., head and neck, trunk, upper extremities, and lower extremities). PASI scores can range from 0.0 to 72.0, with higher scores indicating greater severity and/or more extensive psoriasis.
Percentage of Participants With a Static Physician's Global Assessment (sPGA) Response at Week 4、8、12、16、24、32、48、50 | Week 4、8、12、16、24、32、48、50
  The sPGA is a 6-point scale ranging from 0 (clear) to 5 (very severe) used to measure the severity of disease (induration, scaling, and erythema). A sPGA response is defined as a sPGA value of clear (score 0) or almost clear (score 1).
Change From Baseline in the Percentage of Body Surface Area (BSA) Involved With Psoriasis at Week 4、8、12、16、24、32、48、50 | Baseline and Week 4、8、12、16、24、32、48、50
  A measurement of psoriasis involvement, given as the physician's assessment of the percentage of the participant's total body surface area (BSA) involved with psoriasis. The percent of BSA affected was estimated by assuming that the subject's palm, excluding the fingers and thumb, represented roughly 1% of the body's surface.
  Change from baseline is calculated as (value at post-baseline visit - value at baseline).
  A decrease from baseline (negative value) indicates improvement.
Change From Baseline of dermatology life quality index (DLQI)at Week 4、8、12、16、24、32、48、50 | Baseline and Week 4、8、12、16、24、32、48、50
Positive rate of ADA and NAb | Week1、4、16、32、48、50、52
  Comparision of the positive rate of ADA and NAb between the SCT630 and EU-licensed Humira
Number of Participants With Adverse Events | Week2、4、8、12、16、24、32、40、48、52
Minimum Concentration of SCT630 and EU-licensed Humira | Week1、4、16、32、48、50

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Fourth Military Medical University, Xi'an, Shaanxi, China